CLINICAL TRIAL: NCT05595733
Title: Can Neurally Adjusted Ventilatory Assist Mode Reduce Mechanical Ventilation Day in Patients With Chronic Obstructive Pulmonary Disease ?
Brief Title: Can NAVA Mode Reduce Mechanical Ventilation Day in Patients With COPD ?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fu Jen Catholic University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FJUH110163
Record Dates: First submitted 2022-10-11; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-06

CONDITIONS: Obstructive Lung Diseases
Keywords: Neurally Adjusted Ventilatory Assist; ventilator-free days; patient-ventilator synchrony; diaphragm atrophy; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional group (No Intervention): Using conventional mode to compare mechanical ventilation day with experimental group
- experimental group (Experimental): Using neurally adjusted ventilatory assist mode to compare mechanical ventilation day with conventional group
  Interventions: Device: Ventilator mode

INTERVENTIONS:
Device: Ventilator mode — Neurally Adjusted Ventilatory Assist (NAVA) mode is a new mode of ventilator, using electronic potential of diaphragm to adjust tidal volume. At the same time, this mode can trigger and cycle-off inspiratory time by high sensitivity of electronic potential of diaphragm, increase patient-ventilator synchrony, reduce sedative drug, improve oxygenation, shorten mechanical ventilation day and reduce the rate of diaphragm atrophy. It can improve survival rate and hospital day of patients. Both the animal and human experiment have the effect of lung and diaphragm protection.
  Arms: experimental group

SUMMARY:
Background： Neurally Adjusted Ventilatory Assist (NAVA) mode is a new mode of ventilator, using electronic potential of diaphragm to adjust tidal volume. At the same time, this mode can trigger and cycle-off inspiratory time by high sensitivity of electronic potential of diaphragm, increase patient-ventilator synchrony, reduce sedative drug, improve oxygenation, shorten mechanical ventilation day and reduce the rate of diaphragm atrophy. It can improve survival rate and hospital day of patients. Both the animal and human experiment have the effect of lung and diaphragm protection Effect： The results of this trial are expected to obtain electronic potential of diaphragm in patients with obstructive pulmonary disease. Reviewing the current literature, few related literatures have such data presentation. This trial hopes to evaluate whether the use of NAVA can reduce mechanical ventilation day by analyzing electronic potential of diaphragm in patients with obstructive pulmonary disease.

Investigators expect that participants with obstructive pulmonary disease using NAVA mode will have significantly less mechanical ventilation day than using conventional mode

ELIGIBILITY:
Inclusion Criteria:

1. Obstructive pulmonary diseases include chronic obstructive pulmonary disease (COPD), asthma (Asthma), cystic fibrosis (cystic fibrosis), bronchiectasis (bronchiectasis), bronchiolitis or other diseases that cause airway stenosis, etc.
2. Other patients with obstructive pulmonary disease assessed by the clinical team
3. Consent signed by the principal or legal representative
4. Age > 20 years old and < 99 years old

Exclusion Criteria:

1. Those who cannot place a nasogastric tube due to medical conditions
2. Pregnant women
3. Those who have received gas cutting
4. Patients with phrenic nerve palsy
5. Neuromuscular disease
6. Intubation due to cardiac arrest

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ventilator-free days(VFDs) | up to 28 days
  Each day during the measurement period that participants are both alive and free of mechanical ventilation.
  A participants who is extubated on Day 2 of the study and remains alive and free of the ventilator for the remainder of the 28-day study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Jen Catholic University Hospital All Rights Reserved, Taipei, Taiwan